CLINICAL TRIAL: NCT03739788
Title: Study to Evaluate the Absolute Bioavailability of BMS-986165 Tablet in Healthy Male Participants
Brief Title: An Investigational Study to Evaluate Experimental Medication BMS-986165 Given as a Tablet and Solution in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM011-067; 2018-003134-33 (EudraCT Number)
Record Dates: First submitted 2018-11-09; First posted 2018-11-14 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Healthy Participants
MeSH Terms: interventions — deucravacitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- BMS-986165 (Experimental): Oral and intravenous administration
  Interventions: Drug: BMS-986165

INTERVENTIONS:
Drug: BMS-986165 — Oral administration of tablet and 15-minute intravenous BMS-986165 solution for infusion

SUMMARY:
The purpose of this study is to investigate BMS-986165 given as a tablet in healthy male participants.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy male participant, as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations
* Body mass index (BMI) of 18.0 to 32.0 kg/m2, inclusive, and total body weight ≥ 50 kg (110 lb). BMI = weight (kg)/(height [m])2 at screening
* Normal renal function at screening as evidenced by an estimated glomerular filtration rate (eGFR) ≥ 80 mL/min/1.732

Exclusion Criteria:

* Any medical condition that presents a potential risk to the participant and/or may compromise the objectives of the study, including a history of or active liver disease
* Current or recent (within 3 months of study drug administration) gastrointestinal disease that could impact upon the absorption of study drug
* History or presence of clinically significant acute or chronic bacterial, fungal, or viral infection (eg, pneumonia, septicemia) within the 3 months prior to screening

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
Absolute oral bioavailability (F) of BMS-986165 derived from plasma concentration versus time data | 4 days

SECONDARY OUTCOMES:
Incidence of nonserious adverse events (AE) | Up to 34 days
Incidence of serious adverse events (SAE) | Up to 34 days
Number of clinically significant changes in ECG, vital signs, physical examination findings, or clinical laboratory tests | Up to 34 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm